CLINICAL TRIAL: NCT00001903
Title: Prevention of RSV Infections in Bone Marrow Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990083; 99-I-0083
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Immunization; Immunocompromised; Immunoglobulin; Prophylaxis; Respiratory Virus; Bone Marrow Transplantation; Mini-Transplantation; Peripheral Stem Cell Transplantation
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

INTERVENTIONS:
Drug: RSV Polyclonal Immunoglobulin

SUMMARY:
Respiratory Syncytial Virus (RSV) infections are very common and widespread. By age 5, virtually everyone has been infected and developed antibodies against some strain of the virus. RSV infections happen during adulthood, leading to common cold syndromes. In Bone Marrow Transplant recipients the disease is much more severe, usually progressing to pneumonia. This phenomenon is associated with mortality rates around 60-80%.

RSV Polyclonal Immunoglobulin (Respigam® (Registered Trademark)) has been approved by the Food and Drug Administration and recommended by the American Academy of Pediatrics for prophylaxis of RSV disease in premature babies and children born with bronchopulmonary dysplasia. Furthermore, it has been used to treat RSV pneumonia in children and Bone Marrow Transplant recipients with encouraging results and no complications.

Currently, no preventive strategies are available when approaching this infection among bone marrow transplant patients. We intend to prevent our bone marrow transplant patients from developing RSV pneumonia by employing the strategy already used in premature babies, i.e., by passive immunization with Respigam® (Registered Trademark). Our goal to evaluate the efficacy and safety of this strategy in such immunocompromised population.

We believe that this will be a more reasonable approach than waiting for the infection to settle in and only then treating it, because optimal therapy is not currently available.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) infections are very common and widespread. By age 5, virtually everyone has been infected and developed antibodies against some strain of the virus. RSV infections happen during adulthood, leading to common cold syndromes. In Bone Marrow Transplant recipients the disease is much more severe, usually progressing to pneumonia. This phenomenon is associated with mortality rates around 60-80%.

RSV Polyclonal Immunoglobulin (Respigam® (Registered Trademark)) has been approved by the Food and Drug Administration and recommended by the American Academy of Pediatrics for prophylaxis of RSV disease in premature babies and children born with bronchopulmonary dysplasia. Furthermore, it has been used to treat RSV pneumonia in children and Bone Marrow Transplant recipients with encouraging results and no complications.

Currently, no preventive strategies are available when approaching this infection among bone marrow transplant patients. We intend to prevent our bone marrow transplant patients from developing RSV pneumonia by employing the strategy already used in premature babies, i.e., by passive immunization with Respigam® (Registered Trademark). Our goal to evaluate the efficacy and safety of this strategy in such immunocompromised population.

We believe that this will be a more reasonable approach than waiting for the infection to settle in and only then treating it, because optimal therapy is not currently available.

ELIGIBILITY:
Male or female patients who are between the ages of 2 and 80 years.

Must be admitted to the Bone Marrow Transplant Unit for a bone marrow transplantation (BMT), peripheral stem cell transplantation (PSCT) or mini-transplantation (MT).

Must be in the early phase of BMT, PSCT or MT, i.e., receiving conditioning therapy for the transplant or within the first 30 days of receiving a bone marrow graft or;

Must be greater than 30 days post-engraftment but being treated for Graft vs. Host disease (GVHD) with a total dose of equal to or greater than 1.5 grams/m(2) of methylprednisolone (or equivalent dose of steroids) over the first 3 days.

Must have a negative result (at 48 hours) for RSV in the screening respiratory viral culture.

Less than 8 days have elapsed between meeting eligibility criteria, being contacted by one of the investigators, and making a decision to join the study.

Patients with signs or symptoms of Upper Respiratory Tract infection or pneumonia will be excluded until the etiology is established or RSV is ruled-out by the screening culture.

Patients will be excluded if they have any condition that, in the opinion of the investigator, could affect their safety, preclude evaluation of response, or render unlikely that the contemplated course of therapy can be completed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1999-04; Study Completion 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Whimbey E, Champlin RE, Couch RB, Englund JA, Goodrich JM, Raad I, Przepiorka D, Lewis VA, Mirza N, Yousuf H, Tarrand JJ, Bodey GP. Community respiratory virus infections among hospitalized adult bone marrow transplant recipients. Clin Infect Dis. 1996 May;22(5):778-82. doi: 10.1093/clinids/22.5.778. PMID 8722930
- [Background] Wendt CH, Hertz MI. Respiratory syncytial virus and parainfluenza virus infections in the immunocompromised host. Semin Respir Infect. 1995 Dec;10(4):224-31. PMID 8668850
- [Background] De Vincenzo JP, Leombruno D, Soiffer RJ, Siber GR. Immunotherapy of respiratory syncytial virus pneumonia following bone marrow transplantation. Bone Marrow Transplant. 1996 Jun;17(6):1051-6. PMID 8807113